CLINICAL TRIAL: NCT01494142
Title: Registry for the Atopic Dermatitis Research Network (ADRN-02)
Brief Title: Registry for the Atopic Dermatitis Research Network
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT ADRN-02; NCT00550316 (obsolete NCT alias)
Record Dates: First submitted 2011-10-31; First posted 2011-12-16 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Atopic Dermatitis; Eczema Herpeticum
Keywords: Registry; Atopic Dermatitis; Eczema Herpeticum; GWAS; Staphylococcus aureus
MeSH Terms: conditions — Dermatitis, Atopic; Kaposi Varicelliform Eruption; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood DNA, whole blood RNA,blood cards, blood clots, serum, skin swabs, and skin swab isolates will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- ADEH-Staph+: Atopic Dermatitis without a history of Eczema Herpeticum and with S. aureus skin colonization. A minimum of 1100 participants will be enrolled; we will target 500 Non-Hispanic Caucasian, 300 Non-Hispanic African American, and 300 Mexican American Caucasian ADEH-Staph+ participants. Although we will target these three groups, no racial/ethnic groups will be excluded.
- ADEH-Staph-: Atopic Dermatitis without a history of Eczema Herpeticum and without S. aureus skin colonization. A minimum of 1100 participants will be enrolled; we will target 500 Non-Hispanic Caucasian, 300 Non-Hispanic African American, and 300 Mexican American Caucasian ADEH-Staph- participants. Although we will target these three groups, no racial/ethnic groups will be excluded.
- ADEH+: Atopic Dermatitis with previous or current Eczema Herpeticum.We will try to include a minimum of 150 Non-Hispanic Caucasian ADEH+ participants. ADEH+ participants of other racial/ethnic groups will not be excluded
- ADEV+: Atopic Dermatitis with previous or current Eczema Vaccinatum. ADEV+ sub-phenotype is very rare so all eligible participants will be enrolled.
- Non-atopic: Non-atopic healthy participants. A minimum of 250 non-atopic participants will be enrolled. Non-atopic participants will serve as a control group for the genetic, biomarker, Staph characterization, and microbiome studies.

SUMMARY:
The purpose of this multi-center, clinical registry study is to determine genetic markers associated with susceptibility of AD patients to infections and to also serve as a potential participant database for future studies.

DETAILED DESCRIPTION:
People with atopic dermatitis (AD), also known as eczema, experience hot, dry, scaly skin with severe itching. In addition, people with AD are prone to skin infections and inflammation. Little is known about the causes of AD or why people with AD are more prone to infections. The purpose of this multi-center, clinical registry study is to determine genetic markers associated with susceptibility of AD patients to infections and to also serve as a potential participant database for future studies.

Study procedures will usually be completed in one visit to the clinic; however, participants may need to return for one or more additional visits to provide blood and skin swabs if they do not meet sampling criteria at the initial Screening Visit. A subset of participants from National Jewish Health may be asked to return to clinic for 2 additional visits approximately 7 and 14 days after the original sample collection for collection of skin swabs for assessment of antimicrobial activity. All participants may also be asked to return for an Unscheduled Visit to provide additional blood and/or skin swabs. Atopic Dermatitis with previous or current Eczema Herpeticum (ADEH+), Atopic Dermatitis with previous or current Eczema Vaccinatum (ADEV+) and Methicillin-Resistant S. Aureus (MRSA+) participants will be contacted every 6 months for the duration of the study.

Recruitment emphasis will include Non-Hispanic Caucasian, Non-Hispanic African American, and Mexican American since these constitute the three largest racial/ethnic populations according to the U.S. Census Bureau 2009 data; however, no racial/ethnic groups will be excluded. Our scientific rationale for targeting these three racial/ethnic groups is to ensure that we are able to recruit sufficient numbers of participants in each group to perform meaningful tests for genetic association.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria are eligible for enrollment. Participants may be reassessed if not initially eligible.

* ADEH+ and Non-atopic males and females ages 8 months to 80 years, inclusive, at the time of Enrollment, and ADEH- males and females ages 3 years to 80 years, inclusive, at the time of Enrollment.
* Who are willing to sign the informed consent form or whose parent or legal guardian is willing to sign the informed consent form (age appropriate) prior to initiation of any study procedures.
* Who are willing to sign the assent form, if age appropriate.
* Who meet criteria for one of the diagnostic groups (ADEH-Staph+, ADEH-Staph-, ADEH+, ADEV+, Non-atopic) as defined in the ADRN Standard Diagnostic Criteria and the Staphylococcus aureus Colonization Criteria.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for enrollment.

* Who have an active systemic malignancy; uncomplicated non-melanoma skin cancer and melanoma in situ with documentation of complete excision are not exclusionary.
* Who have any skin disease other than AD that might compromise the stratum corneum barrier (e.g., bullous diseases, psoriasis, cutaneous T cell lymphoma [also called Mycosis Fungoides or Sezary syndrome], dermatitis herpetiformis, Hailey-Hailey, or Darier's disease).
* Who have a history of systemic immunological illness (e.g., immunodeficiency disorders such as human immunodeficiency virus [HIV] or lupus erythematosus) other than the condition being studied.
* Who have a first degree relative already enrolled in the study.
* Who are determined not to be eligible in the opinion of the Investigator.

Ages: 8 Months to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A minimum of 1100 ADEH-Staph+ participants and a minimum of 1100 ADEH-Staph- participants 3-80 years of age will be enrolled. In addition, ADEH+, ADEV+, and Non-atopic participants 8 months to 80 years of age will be enrolled.
  It is unknown whether Staph colonization status will change as younger participants get older. For this reason, the lower age limit for inclusion of ADEH- participants is 3 years rather than 8 months to ensure that characterization of their Staph+ vs. Staph- state is more accurate
Sampling Method: Non-Probability Sample
Enrollment: 3387 (Actual)
Dates: Start 2011-08; Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Genotype and sequence data from ADEH+ and ADEH- participants. | Day 1
Genotype and sequence data from ADEH- participants with and without bacterial colonization with S. aureus. | Day 1

SECONDARY OUTCOMES:
Single Nucleotide Polymorphism (SNP) and Copy Number Variant (CNV) genotype data for candidate genes, including but not limited to Claudin-1 (CLDN1) and Filaggrin (FLG). | Day 1
SNP genotype data for candidate genes, including but not limited to CLDN1 and FLG, validated in samples from an independent AD population. | Day 1
Targeted deep resequencing of candidate genes, including but not limited to CLDN1. | Day 1
Analysis of S. aureus isolates for antibiotic sensitivity | Day 1
Analysis of S. aureus isolates for staphylococcal cassette chromosome (SCC) mec DNA elements. | Day 1
Analysis of S. aureus isolates for expression of virulence or other factors. | Day 1
Expression of biomarkers, including but not limited to serum biomarkers, among AD sub-phenotypes. | Day 1
Analysis of microbial composition by 16S ribosomal Deoxyribonucleic Acid (rDNA) amplicon sequencing. | Day 1
Analysis of DNA methylation profiles | Day 1
Analysis of messenger Ribonucleic Acid (mRNA) expression profiles in whole blood samples. | Day 1
Frequency of commensal Staphylococcus species producing antimicrobial activity | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Beck, MD, Study Chair — University of Rochester; Kathleen Barnes, PhD, Study Chair — Johns Hopkins Asthma and Allergy Center
Locations (9):
- United States (9):
  - Children's Hospital Los Angeles, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Gao L, Bin L, Rafaels NM, Huang L, Potee J, Ruczinski I, Beaty TH, Paller AS, Schneider LC, Gallo R, Hanifin JM, Beck LA, Geha RS, Mathias RA, Barnes KC, Leung DYM. Targeted deep sequencing identifies rare loss-of-function variants in IFNGR1 for risk of atopic dermatitis complicated by eczema herpeticum. J Allergy Clin Immunol. 2015 Dec;136(6):1591-1600. doi: 10.1016/j.jaci.2015.06.047. Epub 2015 Sep 3. PMID 26343451
- [Result] Shi B, Bangayan NJ, Curd E, Taylor PA, Gallo RL, Leung DYM, Li H. The skin microbiome is different in pediatric versus adult atopic dermatitis. J Allergy Clin Immunol. 2016 Oct;138(4):1233-1236. doi: 10.1016/j.jaci.2016.04.053. Epub 2016 Jun 29. No abstract available. PMID 27474122
- [Result] Nakatsuji T, Chen TH, Two AM, Chun KA, Narala S, Geha RS, Hata TR, Gallo RL. Staphylococcus aureus Exploits Epidermal Barrier Defects in Atopic Dermatitis to Trigger Cytokine Expression. J Invest Dermatol. 2016 Nov;136(11):2192-2200. doi: 10.1016/j.jid.2016.05.127. Epub 2016 Jul 2. PMID 27381887
- [Result] Merriman JA, Mueller EA, Cahill MP, Beck LA, Paller AS, Hanifin JM, Ong PY, Schneider L, Babineau DC, David G, Lockhart A, Artis K, Leung DY, Schlievert PM. Temporal and Racial Differences Associated with Atopic Dermatitis Staphylococcusaureus and Encoded Virulence Factors. mSphere. 2016 Dec 7;1(6):e00295-16. doi: 10.1128/mSphere.00295-16. eCollection 2016 Nov-Dec. PMID 27981233
- [Result] Nakatsuji T, Chen TH, Narala S, Chun KA, Two AM, Yun T, Shafiq F, Kotol PF, Bouslimani A, Melnik AV, Latif H, Kim JN, Lockhart A, Artis K, David G, Taylor P, Streib J, Dorrestein PC, Grier A, Gill SR, Zengler K, Hata TR, Leung DY, Gallo RL. Antimicrobials from human skin commensal bacteria protect against Staphylococcus aureus and are deficient in atopic dermatitis. Sci Transl Med. 2017 Feb 22;9(378):eaah4680. doi: 10.1126/scitranslmed.aah4680. PMID 28228596
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait